CLINICAL TRIAL: NCT00667797
Title: Pharmacoeconomic Outcomes of Levalbuterol and Racemic Albuterol in Inpatients Requiring Nebulization (POLARIS)
Brief Title: Costs & Outcomes of Hospitalization/Treatment With Levalbuterol & Albuterol in Asthma or Chronic Obstructive Pulmonary Disease (COPD) Subjects
Acronym: POLARIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 051-921
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Asthma; COPD
Keywords: Asthma; COPD; chronic emphysema; chronic bronchitis
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): levalbuterol 1.25 mg
  Interventions: Drug: levalbuterol HCl
- 2 (Active Comparator): Racemic albuterol 2.5 mg
  Interventions: Drug: albuterol Sulfate

INTERVENTIONS:
Drug: levalbuterol HCl — Levalbuterol 1.25 mg will be prescribed every 6-8 hours, with standing orders for as needed PRN use. However, the prescribing physician may change the dose, frequency, and/or duration of levalbuterol administration at their discretion.
  Other Names: Xopenex Inhalation Solution
  Arms: 1
Drug: albuterol Sulfate — Racemic albuterol 2.5 mg will be prescribed per the standard of care used in the institution, with standing orders for as needed PRN use. However, the prescribing physician may change the dose, frequency, and/or duration of racemic albuterol administration at their discretion.
  Other Names: Ventolin Inhalation Solution
  Arms: 2

SUMMARY:
An analysis of the costs and outcomes associated with hospitalization and treatment of Levalbuterol versus Racemic Albuterol in subjects with Asthma and COPD.

DETAILED DESCRIPTION:
This was a randomized, open-label study evaluating clinical and pharmacoeconomic outcomes in hospitalized patients with asthma or COPD who have been admitted due to an exacerbation of their disease and required further treatment with a beta2-adrenergic agonist. Approximately 430 patients were randomized and enrolled. Patients were then followed during their hospitalization. Once discharged, patient status was assessed via telephone interview 30 days after discharge. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects must be at least greater than or equal to 18 years of age at the time of consent.
* Subjects must have history of asthma or COPD for at least 6 months prior to hospitalization.
* Subjects must have been hospitalized due to an exacerbation of their disease and required further treatment with a nebulized beta2-adrenergic agonist.
* Subjects must have an oxygen saturation level greater than or equal to 90% with greater than or equal to 40% face mask supplemental oxygen.

Exclusion Criteria:

* Subjects who are likely to be in the Intensive Care Unit (ICU) or Critical Care Unit (CCU).
* Based upon history or physical exam in the ED or Clinic, subjects with known or suspected cause of pulmonary symptoms other than asthma or COPD, such as pneumonia, pulmonary embolism, cystic fibrosis, or angioedema. Subjects with CHF that are admitted with a primary admission diagnosis of COPD are not excluded.
* Female subjects who are pregnant or breast feeding.
* Subjects who have participated in an investigational drug study within 30 days of study entry or have previously participated in the current trial.
* Subjects who are planning to receive elective surgical procedures during the 30 day period after hospital discharge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2003-03; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the number of nebulizations, scheduled and rescue, required to treat the patient. | Daily for 14 days

SECONDARY OUTCOMES:
Hospital Length of Stay | Daily for 14 days
Relapse Rate | Daily for 14 days
Clinical Chest Assessment | Daily for 14 days
Pulmonary Function Test Data (FEV1, FVC, PEF, FEV1/FVC) | Pre-dose each day and within 30 minutes after the initial dose of study medication on the first day
Disease Symptoms | Daily for 14 days
Investigator and Subject Global Assessments | Daily for 14 days
Discharge Location Classification | Daily for 14 days
Concomitant Respiratory Medication Use | Daily and 30 days post discharge
Total Hospital Costs | Daily for 14 days
Cost of Respiratory Therapy Resources | Daily for 14 days
Respiratory Medication Costs | Daily for 14 days
Subject Satisfaction with Treatment | Daily for 14 days
Subject General Well-being | Daily and 30 days post discharge

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Birmingham, Alabama
  - Chula Vista, California
  - Oakland, California
  - Wheat Ridge, Colorado
  - Waterbury, Connecticut
  - Washington D.C., District of Columbia
  - Brandon, Florida
  - Des Moines, Iowa
  - Johnson City, New Jersey
  - Great Neck, New York
  - Syracuse, New York
  - Chapel Hill, North Carolina
  - Winston-Salem, North Carolina
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Houston, Texas
  - San Antonio, Texas
  - Morgantown, West Virginia